CLINICAL TRIAL: NCT03046381
Title: A Pilot Open-label Study to Assess the Efficacy and Safety of Tocilizumab in Patients With Active Schnitzler's Syndrome
Brief Title: Tocilizumab in Patients With Schnitzler's Syndrome
Acronym: TOCISCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karoline Krause (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Karoline Krause, Principal Investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOCISCH
Record Dates: First submitted 2017-01-05; First posted 2017-02-08 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Schnitzler's Syndrome
MeSH Terms: conditions — Schnitzler Syndrome | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Other): Tocilizumab 162mg 1x weekly as subcutaneous syringe
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 162mg 1x weekly s.c.
  Other Names: RoActemra®

SUMMARY:
Schnitzler's Syndrome (SchS) is a late-onset multifactorial autoinflammatory disease characterized by chronic urticarial skin lesions and a monoclonal gammopathy usually belonging to the immunoglobulin M (IgM) or IgG class. Symptoms associated with SchS are recurrent fever attacks, bone and muscle pain, arthralgia or arthritis, fatigue and lymphadenopathy. SchS is a rare disease with approximately 300 cases reported in the literature. The nature of SchS is chronic without known reports about spontaneous remissions. Disease onset occurs around the age of 50. About 15% of patients eventually develop a lymphoproliferative disorder, most often Waldenström's macroglobulinemia. The pathogenesis of SchS is still not well defined. Functional ex vivo studies showed excessive cytokine production (IL-1ß, IL-6 and IL-18) of peripheral blood monocytes (PBMCs) in SchS as compared to healthy controls. In addition to excessive IL-6 secretion from PBMCs IL-6 has repeatedly been reported to be elevated in the serum of SchS patients too. As IL-6 plays a major role in the development of multiple myeloma, IL-6 may also be associated with the formation of lymphoproliferative disorders in SchS.

Until now, there is no approved standard therapy available for the treatment of SchS. Non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids, and other immunosuppressive agents have been reported to provide variable relief from symptoms of bone pain and arthralgia. Case reports and small studies about successful treatment of SchS with anti-IL-1 blockers (anakinra, rilonacept and canakinumab) accumulate. However, there have been complete and partial treatment failures to anti-IL-1 blockade in SchS. In these patients, anti-IL-6 treatment (tocilizumab [TCZ]) demonstrated to be very effective in reducing the clinical symptoms and inflammation markers in SchS. TCZ treatment has proved to be very effective, well-tolerated and safe in other acquired autoinflammatory disorders, systemic juvenile idiopathic arthritis (sJIA) and adult-onset Still's disease that share many clinical features (rash, fever, joint involvement, lymphadenopathy, fatigue) and excessive cytokine production with SchS. The study consists of a run-in baseline period of 1-4 weeks followed by an open-label 20-week TCZ treatment phase with weekly s.c. injections (TCZ 162mg), followed by an optional study extension up to a total of 1 year with ongoing once weekly TCZ 162mg injections and a 4 week period of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* SchS diagnosis based on Strasbourg clinical criteria
* Active SchS, refractory to treatment with antihistamines, NSAIDS or colchicine, hydroxychloroquine or dapsone
* Patients who have a symptom score (PGA) of at least 8 (0-20) at baseline
* If necessary, concurrent/ongoing treatment with a stable dose of systemic corticosteroids not greater than 10mg/d for 14 days prior to screening
* If necessary, concurrent/ongoing treatment with a stable dose of antihistamines and NSAIDs for 7 days prior to screening
* Able to read, understand and willing to sign the informed consent form and abide with study procedures
* Willing, committed and able to return for all clinic visits and complete all study-related procedures, including willingness to have SC injections administered by a qualified person
* In females of childbearing potential: Negative pregnancy test within 28 days of randomization; males and females willing to use highly effective contraception (Pearl-Index < 1) during study treatment and for a minimum of 3 months after last dose of TCZ. Pregnancies occurring up to 90 days after the completion of the study medication must be reported to the investigator. A woman will be considered not of childbearing potential if she is post-menopausal for greater than two years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)
* Subjects are considered eligible, if they meet the following tuberculosis (TB) screening criteria: no history of latent or active TB prior to screening, no signs or symptoms suggestive of active TB, no recent close contacts with a person with active TB, and negative QuantiFERON-TB test at screening (if QuantiFERON-TB test is positive, the patient can only be included if active TB is ruled out with appropriate measurements according to standard of care, e.g. the patient is pre-treated with isoniazide for 4 weeks).
* No participation in other clinical trials 4 weeks before and after participation in this study

Exclusion criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Concurrent/ongoing treatment with biologics or recent treatment (less than 5 half lives)

  * With Anakinra within 7 days prior to screening, with canakinumab within 100 days prior to screening
  * with oral/parental corticosteriods greater than 10 mg/d within 2 weeks prior to screening
  * with Cyclosporin A Methotrexate, Dapsone, Chloroquine, Hydroxychloroquine, Azathioprine, Cyclophosphamide within 4 weeks prior to screening
  * other immunosuppressives within 4 weeks or 5 half lives prior to screening, whichever is longer
  * Previous treatment within six months of randomization with any cell-depleting therapies, including investigational agents or approved therapies, some examples include: CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20.
  * Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
* Treatment with a live (attenuated) virus vaccine within 4 weeks prior to Baseline visit
* Significant medical condition rendering the patient immunocompromised or not suitable for a clinical trial
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* An abnormal chest radiograph consistent with clinical signs of prior or present tuberculosis infection whether or not previously treated with anti-tuberculosis agents
* Significant concomitant illness such as, but not limited to, cardiac, renal, neurological, endocrinological, metabolic, or lymphatic disease that would adversely affect the subject's participation or evaluation in this study
* Evidence of current HIV, Hepatitis B, or Hepatitis C infection by clinical or serological history
* Presence of any of the following laboratory abnormalities at enrollment visit: serum creatinine > 1.6 mg/dL (141 µmol/L) in female patients and > 1.9 mg/dL (168 µmol/L) in male patients, WBC <3,000/µl; platelet count <100000/µl ; ALT or AST >2 x ULN or total bilirubin >ULN, Hemoglobin <8.0 g/dL, neutrophil count <2,000 cells/µl or lymphocyte count <500/ µl
* Evidence of active, recurrent or latent systemic infection
* Active systemic inflammatory condition other than SchS including, but not limited to, rheumatoid arthritis
* History of malignancies within five years prior to screening other than a successfully treated non-metastatic cutaneous, basal, or squamous cell carcinoma and/or in situ cervical cancer
* Lactating females or pregnant females
* Enrollment in another investigational treatment or device study or use of an investigational agent, or less than 4 weeks or 5 half-lives, whichever is longer, since end of another investigational device or drug trial
* Subjects for whom there is concern about compliance with the protocol procedures
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk
* History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures.
* Patients with known hypersensitivity to tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Physician global assessment | Baseline vs. week 20
  Change in the investigator's assessment of total disease activity (physician global assessment [PGA]) between baseline and TCZ Treatment

SECONDARY OUTCOMES:
Complete responders | Week 20
  Proportion of patients with complete response (based on PGA with no or minimal overall autoinflammatory disease activity and CRP </= 10 mg/l)
Schnitzler Activity Score | 60 weeks
  Change in the patient based Schnitzler Activity Score (SchAS) during the treatment period (The SchAS combines the key symptoms of SchS).
Inflammation marker CRP | 60 weeks
  Change in CRP levels during the treatment period
Inflammation marker SAA | 60 weeks
  Change in SAA levels during the treatment period
Inflammation marker S100 A8/9 | 60 weeks
  Change in S100 A8/9 levels during the treatment period
Overall quality of life | 60 weeks
  Change in the patient's quality of life (assessed by the SF-36)
Dermatology-specific quality of life | 60 weeks
  Change in the patient's quality of life (assessed by the Dermatology Life Quality Index)
Safety and tolerability assessed by adverse event reporting over the whole study period | 60 weeks
  Adverse event reporting over the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Karoline Krause, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Dpt. of Dermatology and Allergy, Berlin, Germay, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bonnekoh H, Frischbutter S, Roll S, Maurer M, Krause K. Tocilizumab treatment in patients with Schnitzler syndrome: An open-label study. J Allergy Clin Immunol Pract. 2021 Jun;9(6):2486-2489.e4. doi: 10.1016/j.jaip.2021.01.024. Epub 2021 Feb 2. No abstract available. PMID 33545397